CLINICAL TRIAL: NCT04644133
Title: Assessment of Daily Electronic Stool Diary for Constipation and Fecal Incontinence.
Brief Title: Electronic Mobile Phone App Stool Diary
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Satish Rao, Professor, Augusta University
Other Study IDs: 1297973
Record Dates: First submitted 2020-07-31; First posted 2020-11-25 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Constipation; Incontinence Bowel
MeSH Terms: conditions — Constipation; Encopresis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy: Subjects without bowel issues will be asked to complete a 2 week electronic stool diary and a 2 week paper stool diary. They will complete feedback questionnaires for comparison between the two forms of diaries. The subjects will have the option to download the Stool Dairy App or if they do not have access to a smartphone they will be provided with a phone on which one the app has already been uploaded and instructed on its use. Subject's charts may be reviewed.
  Interventions: Other: Paper diary; Other: Electronic APP diary
- Constipation: Subjects diagnosed with constipation will be asked to complete a 2 week electronic stool diary and a 2 week paper stool diary. They will complete feedback questionnaires for comparison between the two forms of diaries. The subjects will have the option to download the Stool Dairy App or if they do not have access to a smartphone they will be provided with a phone on which one the app has already been uploaded and instructed on its use. Subject's charts may be reviewed.
  Interventions: Other: Paper diary; Other: Electronic APP diary
- Fecal Incontinence: Subjects diagnosed with fecal incontinence will be asked to complete a 2 week electronic stool diary and a 2 week paper stool diary. They will complete feedback questionnaires for comparison between the two forms of diaries. The subjects will have the option to download the Stool Dairy App or if they do not have access to a smartphone they will be provided with a phone on which one the app has already been uploaded and instructed on its use. Subject's charts may be reviewed.
  Interventions: Other: Paper diary; Other: Electronic APP diary

INTERVENTIONS:
Other: Paper diary — Subjects will be asked to complete a 2 week paper stool diary.
Other: Electronic APP diary — Subjects will be asked to complete a 2 week paper stool diary.

SUMMARY:
Our objective here is to improve the patient's compliance and accurate capture of patient reported bowel and abdominal symptoms, by utilizing a phone application that interactively records each bowel movement or leakage event and other bowel symptoms. Such an electronic stool diary may relieve the burden of using a paper daily stool diary. We will compare and validate the electronic stool diary with the paper stool diary.

DETAILED DESCRIPTION:
Fecal incontinence consists of multiple and often unpredictable bowel movements and leakage of stool. Chronic constipation is associated with episodes of irregular and unpredictable bowel habits and difficulty with remembering symptoms. These features lead to a recall bias, and inaccurate recollection and/or documentation of symptoms that are critical for diagnosis and management. A daily stool diary has been used in clinical trials and in clinical practice to accurately record bowel symptoms. However, patients find these diary entries cumbersome or embarrassing to use, especially with bowel movements that occur outside of home resulting in loss of data or inaccurate collection of information. Also, many patients forget events especially when this bowel habit is irregular. Therefore, it is crucial to explore new ways of accurately, reliability, and more discretely collect bowel habit information, by using current technology that a majority of people have access to.

ELIGIBILITY:
Inclusion Criteria:

* Anyone older than 18 years with symptoms of Fecal Incontinence (FI), Constipation, or Healthy (i.e. no bowel issues).
* Women of childbearing age will be asked if they are pregnant, and a confirmed negative response is given will be sufficient. No pregnancy test will be performed.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Anyone symptoms of Fecal Incontinence (FI), Constipation, or Healthy (i.e. no bowel issues).
Sampling Method: Non-Probability Sample
Enrollment: 135 (Estimated)
Dates: Start 2018-12-06 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Correlation of electronic APP diary information with paper form stool diary in healthy subjects | 2 weeks each
  The stool diary parameters: number of bowel movements, number of leakages, stool consistency, urgency, time spent on toilet, feeling of incomplete evacuation,straining, gas and bloating recorded in the paper form stool diary over 2 weeks will be correlated with the electronic APP stool diary parameters using Pearson correlation in healthy subjects.
Correlation of electronic APP diary information with paper form stool diary in fecal incontinence subjects | 2 weeks each
  The stool diary parameters; number of bowel movements, number of leakages, stool consistency, urgency, sensation before leakage, feeling of incomplete evacuation,use of pads and medication use recorded in the paper form stool diary over 2 weeks will be correlated with the electronic APP stool diary parameters using Pearson correlation in fecal incontinence subjects
The stool diary parameters | 2 weeks each
  The stool diary parameters: number of bowel movements, stool consistency, urgency, time spent on toilet, feeling of incomplete evacuation,straining, gas and bloating recorded in the paper form stool diary over 2 weeks will be correlated with the electronic APP stool diary parameters using Pearson correlation in constipation subjects

SECONDARY OUTCOMES:
Stool frequency | 2 weeks
  The number of bowel movements per week (BM), the number of spontaneous bowel movements (SBM), and the number of complete spontaneous bowel movements (CSBM) will be compared between the APP and stool diary and between healthy subjects and patients with constipation and fecal incontinence.
Stool consistency | 2 weeks
  Stool consistency (Bristol Stool scale, 1-7): 1-very hard stool, 4- normal, smooth stool, 7- watery stool, will be compared between the APP and stool diary and between healthy subjects and patients with constipation and fecal incontinence.
Bowel urgency | 2 weeks
  Severity of bowel urgency- unable to postpone BM for more than 15 minutes, will be compared between the APP and stool diary and between healthy subjects and patients with constipation and fecal incontinence.
Stool leakage | 2 weeks
  Leakage characteristics-amount: 0- none, 1-mild, 2-moderate, 3- excessive, will be compared between the APP and stool diary and between healthy subjects and patients with fecal incontinence.
Complete evacuation | 2 weeks
  Feeling of complete evacuation, will be compared between the APP and stool diary and between healthy subjects and patients with constipation and fecal incontinence.
Week 1 vs Week 2 reproducibility of APP and paper diary | 1 weeks
  Compare the results for the first and the second week for the electronic APP data as well as paper data and examine the reproducibility.
Straining | 2 weeks
  Stool straining will be compared between the APP and stool diary and between healthy subjects and patients with constipation.
Time spent of toilet | 2 weeks
  Time spent on toilet will be compared between the APP and stool diary and between healthy subjects and patients with constipation.

CONTACTS AND LOCATIONS:
Overall Officials: Satish Rao, MD PhD, Study Director — Augusta University
Locations (1):
- Digestive Health Clinical Research, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided